CLINICAL TRIAL: NCT01217528
Title: Reduction of Inappropriate ICD Therapies in Patients With Approved Indication for Primary Prevention of Sudden Cardiac Death
Brief Title: Reduction of Inappropriate Implantable Cardioverter Defibrillator (ICD) Therapies in Primary Prevention Patients
Acronym: DECREASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T76
Record Dates: First submitted 2010-09-10; First posted 2010-10-08 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Death
Keywords: ICD; CRTD; Sudden cardiac death; Device settings; Patients who received ICD/CRTD for primary prevention of sudden cardiac death
MeSH Terms: conditions — Death; Death, Sudden, Cardiac | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Group A:
  * VT zone: 350ms
  * VF zone: 280ms
  Interventions: Device: device settings for group A
- Group B (Experimental): Group B:
  * VT zone: 320ms
  * VF zone: 250ms
  Interventions: Device: Device settings for group B

INTERVENTIONS:
Device: device settings for group A — VT zone: 350ms VF zone: 280ms
  Other Names: Control group
  Arms: Group A
Device: Device settings for group B — VT zone: 320ms VF zone: 250ms
  Other Names: Treatment group
  Arms: Group B

SUMMARY:
The purpose of this study is to determine efficacy of a dedicated programming concept for avoidance of inappropriate implantable cardioverter defibrillator (ICD) therapies in patient with primary prevention ICD indication.

DETAILED DESCRIPTION:
Inappropriate ICD therapies still remains a major issue with respect to patient's quality of life and proarrhythmic risk.

It's the aim of this study to determine efficacy of a dedicated programming concept for avoidance of inappropriate ICD therapy in patients who received the ICD for primary prevention of sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

* Approved indication for new ICD implantation for primary prevention of sudden cardiac death
* Age >=18 Years
* Written informed consent

Exclusion Criteria:

* ICD indication for secondary prevention reasons
* ICD indication for "electrical" disorders (i.e. long/short QT syndrome, Brugada syndrome etc...)
* ICD change or upgrade
* Pregnancy
* Nonage
* Patient is already participating to another study with active therapy arm
* Patient will most likely not be able to participate to the routine follow ups in the study center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2009-08; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 12 months
  Event free survival of:
  1. inappropriate ICD therapies (only stored tachycardias with proper stored EGM documentation are taken into account) AND
  2. spontaneous, documented, sustained (>30s) ventricular tachycardia, that was not treated by the ICD

SECONDARY OUTCOMES:
Amount of patients with appropriate / inappropriate ICD therapies | 12 months
Prevalence of slow VT (<=187bpm) in patients with indication for primary prevention of SCD | 12 months
Number and cycle lengths of supraventricular / ventricular tachys | 12 months
Time to first appropriate / inappropriate ICD therapy | 12 months
Sensitivity for diagnosis of sustained VT | 12 months
Specificity for SVT diagnosis | 12 months
Quality of Life (MLHF Questionaire) | 12 months
Overall mortality | 12 months
Cardiac mortality | 12 months
Frequency and efficacy of ATP prior to / before capacitor charging in VF zone | 12 months
Amount of patients with appropriate / inappropriate shocks or ATP | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jörg O Schwab, Prof. Dr. med., Principal Investigator — Medizinische Einrichtungen der Rheinischen Friedrich-Wilhelm-Universität Bonn
Locations (34):
- Germany (34):
  - Medizinische Einrichtungen der RWTH Aachen, Aachen
  - Klinikum Altenburger Land GmbH, Altenburg
  - Städtisches Krankenhaus St. Barbara Attendorn GmbH, Attendorn
  - Medizinische Einrichtungen der Rheinischen Friedrich-Wilhelm-Universität, Bonn
  - Klinikum Coburg, Coburg
  - Evangelisches Krankenhaus Kalk, Cologne
  - Klinik Fränkische Schweiz, Ebermannstadt
  - Kreiskrankenhaus Ebersberg, Ebersberg
  - Kardiologische Gem.-Praxis Dres. med. Bischoff / Lang, Erfurt
  - Klinikum Esslingen, Esslingen am Neckar
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Krankenhaus Waltershausen-Friedrichroda, Friedrichroda
  - Universitätsklinikum Gießen und Marburg GmbH - Standort Gießen, Giessen
  - Asklepios Klinik St. Georg, Hamburg
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Oberhavel Kliniken GmbH Klinik Hennigsdorf, Henningsdorf
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Frankenwaldklinik Kronach GmbH, Kronach
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - St.-Marien-Hospital GmbH, Lünen
  - Klinikum Memmingen, Memmingen
  - Klinikum Großhadern der Ludwig-Maximilians-Universität München, München
  - Herzkatheter / Praxisklinik Dres. med. Mühling / Prof. Dr. Silber, München
  - Universitätsklinikum Münster, Münster
  - Praxis Dres. med. Haggenmiller / Jeserich, Nuremberg
  - Klinikum Nürnberg, Nuremberg
  - Kreiskrankenhaus des Bördekreises Krankenhaus 4, Oschersleben
  - Niels-Stensen-Kliniken Marienhospital Osnabrück, Osnabrück
  - Klinikum Pirna GmbH Klinik für Innere Medizin II, Pirna
  - Klinikum Dorothea Christiane Erxleben GmbH, Quedlinburg
  - Wilhelm-Augusta Krankenhaus des Deutschen Roten Kreuzes, Ratzeburg
  - Universität Rostock, Rostock
  - Katharinen-Hospital gGmbH, Unna
  - Helios Klinikum Wuppertal, Wuppertal

REFERENCES:
- [Derived] Schwab JO, Bonnemeier H, Kleemann T, Brachmann J, Fischer S, Birkenhauer F, Eberhardt F. Reduction of inappropriate ICD therapies in patients with primary prevention of sudden cardiac death: DECREASE study. Clin Res Cardiol. 2015 Dec;104(12):1021-32. doi: 10.1007/s00392-015-0870-z. Epub 2015 May 23. PMID 26002818